CLINICAL TRIAL: NCT04611126
Title: T-cell Therapy in Combination With Nivolumab, Relatlimab and Ipilimumab for Patients With Advanced Ovarian-, Fallopian Tube- and Primary Peritoneal Cancer
Brief Title: T-cell Therapy in Combination With Nivolumab, Relatlimab and Ipilimumab for Patients With Metastatic Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, M.D., Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GY2028
Record Dates: First submitted 2020-10-20; First posted 2020-11-02 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Ovarian Cancer; Metastatic Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Adoptive Cell Therapy; Immune Therapy; Tumor Infiltrating Lymphocytes
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Ipilimumab; Cyclophosphamide; fludarabine phosphate; Nivolumab; relatlimab

STUDY DESIGN:
Intervention Model Description: 18 patients are included in 3 steps, containing 6 patients each.
  Step 1: 6 patients will be included. Ipilimumab wil not be administered pre-tumor harvest. If feasible and tolerable, as defined by no additional SAE/SAR compared to the previously completed pilot studies at CCIT-DK, the trial will move to Step 2
  Step 2: 6 patients will be included. Ipilimumab will be administered once 2-6 weeks before tumor resection.
  Step 3: If no additional SAE/SAR, compared to the previous completed study at CCIT-DK, is observed additional 6 patients can be included at Step Two. If on the other hand Step 2 is not found safe, additional 6 patients can be included at Step 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without Ipilimumab (Other): At Step 1, 6 patients will be treated without Ipilimumab pre tumor harvest. If feasible and tolerable, as defined by no additional SAE/SAR compared to the previously completed pilot studies at CCIT-DK, the trial will move to Step 2.
  Depending on the safety and feasibility on step 2, 6 more patients can be included at step 1.
  Interventions: Drug: Cyclophosphamid; Drug: Fludarabine Phosphate; Biological: Tumor Infiltrating Lymphocytes infusion; Drug: Nivolumab; Drug: Relatlimab
- With Ipilimumab (Other): At Step 2, 6 patients will be included. Ipilimumab 3 mg/kg will be administered 2-6 weeks pre tumor harvest.
  If no additional SAE/SAR compared to the previous completed pilot study at CCIT-DK is observed additional 6 patients can be included at Step 2. If on the other hand Step 2is not found safe additional 6 patients can be included at Step 1
  Interventions: Drug: Ipilimumab; Drug: Cyclophosphamid; Drug: Fludarabine Phosphate; Biological: Tumor Infiltrating Lymphocytes infusion; Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3 mg/kg is administered 2-6 weeks before surgical removement of the tumor. The medicine is administered i.v. over 30 minutes.
  Arms: With Ipilimumab
Drug: Cyclophosphamid — Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Other Names: Cyclophosphamide
Drug: Fludarabine Phosphate — Fludarabine 25 mg/m2 is administered on day -5 to day -1.
Biological: Tumor Infiltrating Lymphocytes infusion — Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion. The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Other Names: TILs
Drug: Nivolumab — Nivolumab 240 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 30 minutes.
Drug: Relatlimab — Relatlimab 80 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 60 minutes.
  Other Names: Relalimab

SUMMARY:
Although immunotherapy has revolutionized the treatment of many cancers, ovarian cancer patients have not yet benefitted from the advances.

In two consecutive pilot trials at National Center for Cancer Immune Therapy (CCIT-DK), is has been have shown that adoptive cell therapy (ACT) with TILs for patients with advanced ovarian cancer (OC) is feasible and tolerable. In the most recent of these trials ACT was combined with a CTLA-4 inhibitor, Ipilimumab and a PD1-inhibitor, Nivolumab. Only transient clinical responses where observed.

Between 90-100 % of infused T-cells in our previous ovarian cancer ACT trial expressed LAG-3. The interaction between LAG-3 on T-cells and MHC-II on tumor cells inhibits T-cell function.

In this study adding the LAG-3 antibody Relatlimab to the ACT-regimen described above may therefore well unleash T-cell antitumor efficacy by blocking the known LAG-3-MHC-II interaction.

With this study the aim is to demonstrate that adding the lag-3-inhibitor Relatlimab to the above treatment regimen is feasible and tolerable. The study will elucidate whether the combination Relatlimab-Nivolumab leads to objective responses and improves progression free survival (PFS).

DETAILED DESCRIPTION:
Rationale T-cell therapy is an experimental personalized immunotherapy where TILs are isolated from the patient's own tumor tissue, expanded in vitro to billions of cells and then administered to the individual patient with the purpose of eliminating the remaining cancer cells. Lymphodepleting chemotherapy with cyclophosphamide and fludarabine phosphate is administered to the patient before TIL infusion to reduce the number of irrelevant immune cells.

In two consecutive pilot trials at National Center for Cancer Immune Therapy (CCIT-DK), it has been shown that adoptive cell therapy (ACT) with TILs for patients with advanced ovarian cancer (OC) is feasible and tolerable. In the most recent of these trials ACT was combined with a CTLA-4 inhibitor, Ipilimumab and a PD1-inhibitor, Nivolumab.

Between 90-100% of infused T-cells in these previous ovarian cancer ACT trial expressed LAG-3. The interaction between LAG-3 on T-cells and MHC-II on tumor cells inhibits T-cell function.

In this phase I/II study 18 patients with advanced ovarian -, fallopian tube-, and primary peritoneal cancer will be included. Included patients undergo surgical removal of tumor tissue for tumor-infiltrating lymphocyte (TIL) manufacturing. Lymphodepleting chemotherapy is administered prior to TIL infusion. Hereafter the patients are treated with the programmed cell death protein 1 (PD-1) antibody Nivolumab and the anti-lymphocyte activation gene 3 (anti-LAG-3) antibody Relatlimab. The study will be divided into 3 steps.

* Step One (6 subjects): Patients are treated without prior administration of cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) antibody Ipilimumab pre-tumor harvest.
* Step Two (6 subjects): If Step One proves feasible and tolerable patients in Step Two will receive one dose of Ipilimumab pre-tumor harvest.
* Step Three (6 subjects): Patients are treated either with or without prior Ipilimumab pre-tumor harvest depending on the tolerability data from Step Two.

All patients are treated with lymphodepleting chemotherapy for 7 days followed by infusion of TILs. For safety reasons no IL-2- will be administered in this study

The aim of this study is to demonstrate that ACT and a combination of Relatlimab-Nivolumab does not increase the toxicity compared to the same treatment regimen including Nivolumab monotherapy. The study will elucidate whether the combination Relatlimab-Nivolumab lead to objective responses and improves progression free survival (PFS). It is anticipated that combining Relatlimab and Nivolumab with Adoptive T cell therapy (ACT) for advanced OC is safe and feasible. Further, it is hypothesized that the combination will lead to improved immunity in tumor and blood as well as improved antitumor efficacy.

Objectives

* To evaluate the tolerability and safety of the treatment
* To characterize antitumor immune responses and clinical efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven advanced ovarian-, fallopian tube or primary peritoneal cancer with the possibility of surgical removal of tumor tissue of > 1 cm3. All histologies can be included.
2. Progressive or recurrent resistant disease after platin-based chemotherapy (platinum resistant) or progressive or recurrent disease after second line or additional chemotherapy.
3. Age: 18 - 75 years.
4. ECOG performance status of ≤1 (Appendix 2).
5. Life expectancy of > 6 months.
6. At least one measurable parameter in accordance with RECIST 1.1 -criteria.
7. LVEF assessment with documented LVEF ≥50% by either TTE or MUGA (TTE preferred test) within 6 months from first study drug administration
8. No significant toxicities or side effects (CTC ≤ 1) from previous treatments, except sensory- and motoric neuropathy (CTC ≤ 2) and/or alopecia (CTC ≤ 2).
9. Sufficient organ function, including:

   * Absolute neutrophil count (ANC) ≥ 1.500 /µl
   * Leucocyte count ≥ lower normal limit
   * Platelets ≥ 100.000 /µl and <700.000 /µl
   * Hemoglobin ≥ 6,0 mmol/l (regardless of prior transfusion)
   * S-creatinine < 140
   * S-bilirubin ≤ 1,5 times upper normal limit
   * ASAT/ALAT ≤ 2,5 times upper normal limit
   * Alkaline phosphatase ≤ 5 times upper normal limit
   * Lactate dehydrogenase ≤ 5 times upper normal limit
   * Sufficient coagulation: APPT<40 and INR<1,5
10. Signed statement of consent after receiving oral and written study information
11. Willingness to participate in the planned controls and capable of handling toxicities.
12. Age and Reproductive Status: Females, ages ≥18 years, inclusive

    * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of study treatment.Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception. This applies from inclusion in the study and for the duration of treatment with Ipilimumab, Relatlimab and Nivolumab plus 5 half-lives of study treatment plus 30 days (duration of ovulatory cycle) for a total of 24 weeks post-treatment completion. The following are considered safe methods of contraception:
    * Hormonal anticonception (birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring and transdermal depot patch)
    * Intrauterine device
    * Surgical sterilization
    * Surgical sterilization of male partner with verification of no sperm after the procedure
    * Menopause (for more than 12 months)

Exclusion Criteria:

Patients will be excluded if they meet one of the criteria's listed below

1. A history of prior malignancies. Patients treated for another malignancy can participate if they are without signs of disease for a minimum of 3 years after treatment.
2. Known hypersensitivity to one of the active drugs or one or more of the excipients.
3. Severe medical conditions, such as severe asthma/COLD, significant cardiac disease, poorly regulated insulin dependent diabetes mellitus among others.
4. Creatinine clearance < 70 ml/min (1).
5. Acute/chronic infection with HIV, hepatitis, syphilis among others.
6. Severe allergies or previous anaphylactic reactions.
7. Active autoimmune disease, such as autoimmune neutropenia/thrombocytopenia or hemolytic anemia, systemic lupus erythematosis, Sjögren's syndrome, sclerodermia, myasthenia gravis, Goodpasteur's disease, Addison's disease, Hashimotos thyroiditis, active Graves disease.
8. Subjects with history of myocarditis, regardless of etiology
9. Troponin T (TnT) or I (TnI) > 2x institutional upper limit of normal (ULN) is excluded. ii) between > 1 to 2 x ULN will be permitted if a repeat assessment remains ≤ 2 x ULN and participant undergoes a cardiac evaluation and is cleared by a cardiologist or cardio-oncologist
10. Prior treatment with LAG-3 targeted agents.
11. Pregnant women and women breastfeeding.
12. Simultaneous treatment with systemic immunosuppressive drugs (including prednisolone, methotrexate among others) (2).
13. Simultaneous treatment with other experimental drugs. Based on clinical judgement antihormonal treatment can be accepted.
14. Simultaneous treatment with other systemic anti-cancer treatments.
15. Patients with active and uncontrollable hypercalcemia

(1)In selected cases it can be decided to include a patient with a GFR < 70 ml/min with the use of a reduced dose of chemotherapy.

(2)In selected cases a systemic dose of ≤10 mg prednisolone or a transient planned treatment that can be stopped before TIL therapy can be tolerated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof., M.D., Study Director — Study Director, National Center for Cancer Immune Therapy, Dept. of Oncology, Hospital Herlev; Tine J Monberg, M.D., Study Director — Clinical Assistant, National Center for Cancer Immune Therapy, Dept. of Oncology, Hospital Herlev
Locations (1):
- National Center for Cancer Immune Therapy (CCIT-DK), Herlev, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Without Ipilimumab: At Step 1 the patients received:
  Cyclophosphamid: Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Fludarabine Phosphate: Fludarabine 25 mg/m2 is administered on day -5 to day -1.
  Tumor Infiltrating Lymphocytes infusion: Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion. The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Nivolumab: Nivolumab 240 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 30 minutes.
  Relatlimab: Relatlimab 80 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 60 minutes.
  Due to the premature closure of the trial only 6 patients were enrolled.
- With Ipilimumab: The trial was prematurely closed before step 2
Period: Overall Study
Arm/Group | Without Ipilimumab | With Ipilimumab
Started | 6 (Initially, inclusion of 18 patients in three steps was planned. However, due to the premature closure of the trial, only 6 patients were enrolled.) | 0
Completed | 5 | 0
Not Completed | 1 | 0
Not completed — TIL expansion unsuccessful | 1 | 0

BASELINE CHARACTERISTICS:
Population: As stated in the "Participant Flow", Six patient were enrolled in the trial. However, due to TIL expansion failure one patient was excluded and did never received any treatment in the protocol. Thus, the analysis is performed on the 5 patients that were actually treated in the protocol.
  Due to the premature closure of the trial, no patients were ever included in step two (with ipilimumab) and the expected number of participant (18) was never reached.
Groups:
- Without Ipilimumab: At Step one, 6 patients were enrolled. Due to one expansion failure 5 patients were treated with:
  Cyclophosphamid: Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Fludarabine Phosphate: Fludarabine 25 mg/m2 is administered on day -5 to day -1.
  Tumor Infiltrating Lymphocytes infusion: Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion. The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Nivolumab: Nivolumab 240 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 30 minutes.
  Relatlimab: Relatlimab 80 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 60 minutes.
- With Ipilimumab: This step never started due to slow recruitment
- Total: Total of all reporting groups
Arm/Group | Without Ipilimumab | With Ipilimumab | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 2 |  | 2
Age, Continuous [Median (Full Range); unit: years] | 62 [45 to 70] |  | 62 [45 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 5 |  | 5
Histology [Number; unit: participants]
  High grade serous adenocarcinoma assessed by trained pathologist | 2 |  | 2
  Low grade serous adenocarcinoma assessed by trained pathologist | 2 |  | 2
  Undifferentiated carcinoma assessed by trained pathologist | 1 |  | 1
Number of prior treatment lines [Median (Full Range); unit: lines] | 3 [3 to 4] |  | 3 [3 to 4]
Performance status assessed by the ECOG Performance Status Scale [Count of Participants; unit: Participants] — ECOG Performance status:
  0: Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair
  ECOG PS grade 0-1 was required for inclusion in the trial
  Participants
    ECOG PS 0 | 3 |  | 3
    ECOG PS 1 | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Excluded Due to Treatment Related Safety Issues
Description: Number of patients excluded due to treatment related safety issues compared to the number of patients enrolled in the study
Time Frame: Until completion of the study for
Population: The trial was prematurely closed due to slow patient recruitment. Thus, step 2 was never started.
Measure: Count of Participants; unit: Participants
Groups:
- Without Ipilimumab: At Step 1, 5 patients were treated with:
  Cyclophosphamid: Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Fludarabine Phosphate: Fludarabine 25 mg/m2 is administered on day -5 to day -1.
  Tumor Infiltrating Lymphocytes infusion: Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion. The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Nivolumab: Nivolumab 240 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 30 minutes.
  Relatlimab: Relatlimab 80 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 60 minutes.
- With Ipilimumab: The trial was prematurely closed due to slow recruitment.
Arm/Group | Without Ipilimumab | With Ipilimumab
Number analyzed (Participants) | 6 | 0
Participants | 0 | 0

2. Primary Outcome: Number of Participants Experiencing Grade III or Worse Adverse Events
Description: The number of Participants Experiencing Grade III or Worse Adverse Events
Time Frame: Until completion of the study
Population: The trial was prematurely closed due to slow patient recruitment. Thus, step 2 was never started.
Measure: Count of Participants; unit: Participants
Groups:
- Without Ipilimumab: At Step 1, 5 patients were be treated with
  Cyclophosphamid: Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Fludarabine Phosphate: Fludarabine 25 mg/m2 is administered on day -5 to day -1.
  Tumor Infiltrating Lymphocytes infusion: Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion. The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Nivolumab: Nivolumab 240 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 30 minutes.
  Relatlimab: Relatlimab 80 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 60 minutes.
- With Ipilimumab: The trial was prematurely closed due to slow patient recruitment. Thus, step 2 was never started.
Arm/Group | Without Ipilimumab | With Ipilimumab
Number analyzed (Participants) | 5 | 0
Participants
  Number of Participants Experiencing Grade III or Worse Adverse Events | 5 | 0
  Number of Participants with no Grade III or Worse Adverse Events | 0 | 0

3. Primary Outcome: Number of Patients Excluded Due to Feasibility Issues
Description: Number of patients excluded due to feasibility issues compared to the number of patients enrolled in the study
Time Frame: Until completion of the study
Population: The trial was prematurely closed due to slow patient recruitment. Thus, step 2 was never started.
Measure: Count of Participants; unit: Participants
Groups:
- Without Ipilimumab: A total of six patients were enrolled in the trial
Arm/Group | Without Ipilimumab | With Ipilimumab
Number analyzed (Participants) | 6 | 0
Participants | 1 | 0

4. Secondary Outcome: Best Overall Response (BOR)
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) assessed by CT scan. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions Overall Response (OR) = CR + PR.
Time Frame: The patients were evaluated every 6-12 weeks after therapy and until study completion
Population: The trial was prematurely closed due to slow patient recruitment. Thus, step 2 was never started.
Measure: Count of Participants; unit: Participants
Groups:
- Without Ipilimumab: At Step 1, 5 patients were treated with
  Cyclophosphamid: Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Fludarabine Phosphate: Fludarabine 25 mg/m2 is administered on day -5 to day -1.
  Tumor Infiltrating Lymphocytes infusion: Tumor-infiltrating lymphocytes grown ex-vivo from resected from cancer tissue and reapplied to the patient via an intravenous infusion. The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Nivolumab: Nivolumab 240 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 30 minutes.
  Relatlimab: Relatlimab 80 mg i.v. is administered on day -2 and every 2 weeks for a total of 4 doses. The medicine is administered over 60 minutes.
Arm/Group | Without Ipilimumab | With Ipilimumab
Number analyzed (Participants) | 5 | 0
Participants
  Stable disease | 3 | 0
  Unconfirmed partial response | 2 | 0

ADVERSE EVENTS:
Time Frame: The data was collected throughout the duration of the clinical trial. From April 2021 (enrollment of the first patient) and until exclusion of the last patient in March 2024 (2 years, 11 months) For the individual patient, the reporting started at study enrolment and ended with study exclusion (minimum of 6 months follow-up after therapy or until study completion), up to 9.5 months Adverse events were collected every 6 weeks for the first 3 months and every 3 months hereafter, median 92 days.
Description: Serious adverse events also includes AEs that
  * results in persistent or significant disability or incapacity;
  * leads to a congenital anomaly or birth defect;
  * is a significant medical event.
  * results in the transmission of an infectious agent
  * pregnancy must follow the same transmission timing and process used for SAEs.
  A specific list of events that should not be reported is included in the protocol
Arm/Group | Without Ipilimumab | With Ipilimumab
All-Cause Mortality (participants affected / at risk) | 4/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/5 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Without Ipilimumab (N=5) | With Ipilimumab (N=0)
Bacterial infection (Infections and infestations) | 1 (1) | 0
Ileus (small intestine) (Gastrointestinal disorders) | 1 (1) | 0 — Ileus, presumably caused by carcinosis
Atrial febrillation (Cardiac disorders) | 1 (1) | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Colon ileus (Gastrointestinal disorders) | 1 (1) | 0 — Due to carcinosis and/or infection with clostridium difficile
Gastroenteritis (Gastrointestinal disorders) | 1 (2) | 0
Kidney failure (General disorders) | 1 (1) | 0 — Kidney failure secondary to colon ileus and infection
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 — Cardiac effusion caused by pericardial metastases
Hyperthyroidism (Endocrine disorders) | 1 (2) | 0
Bacterial infection during neutropenia (Infections and infestations) | 1 (1) | 0
Reactivation of Cytomegalo virus (Infections and infestations) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Without Ipilimumab (N=5) | With Ipilimumab (N=0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 0
Neutropenia (Blood and lymphatic system disorders) | 5 (8) | 0
Anemia (Blood and lymphatic system disorders) | 5 (7) | 0
Hyponetriemia (Blood and lymphatic system disorders) | 5 (7) | 0
Nausea (Gastrointestinal disorders) | 5 (6) | 0
Trombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 0
Decrease in PS (General disorders) | 5 (9) | 0
Fatique (General disorders) | 5 (9) | 0
Infections (Infections and infestations) | 3 (7) | 0
Vomiting (Gastrointestinal disorders) | 3 (3) | 0
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0
Obstipation (Gastrointestinal disorders) | 2 (2) | 0
Dry mouth (Gastrointestinal disorders) | 2 (4) | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Elevated ALAT/ASAT (Hepatobiliary disorders) | 2 (2) | 0
Increased p-ferritin (Blood and lymphatic system disorders) | 1 (1) | 0
Oral candida (Infections and infestations) | 1 (2) | 0
Fever (General disorders) | 4 (7) | 0
Maculopapular rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0
Troponine increase (Cardiac disorders) | 1 (2) | 0
Increased ferritin (Blood and lymphatic system disorders) | 1 (1) | NA
Elevated creatinine (Renal and urinary disorders) | 1 (1) | NA
Hyperthyroidism (Endocrine disorders) | 2 (2) | NA
Obstipation (Gastrointestinal disorders) | 3 (3) | NA
Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | NA

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT04611126/Prot_SAP_000.pdf